CLINICAL TRIAL: NCT07202468
Title: "The Effect of Two Different Applications Shown With Virtual Reality Glasses During Peripheral Venous Catheterization on Pain, Fear, and Physiological Parameters in Children"
Brief Title: Virtual Reality for Pain, Fear, and Physiological Responses During Pediatric Venous Catheterization
Acronym: VR-PainKids
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Burak Genç, Research Assistant, Ege University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 1051
Record Dates: First submitted 2025-09-12; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Pain Management; Fear and Anxiety
MeSH Terms: conditions — Agnosia; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Children were randomly assigned into three parallel groups: (1) Aquarium VR intervention, (2) Kaleidoscope VR intervention, and (3) routine care control group. Outcomes were compared across groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aquarium VR intervention group (Experimental): Children wore a virtual reality headset displaying a 3D aquarium video with underwater scenes. The headset was applied 2-3 minutes before peripheral intravenous catheterization and continued during the procedure to provide distraction.
  Interventions: Device: Virtual Reality
- Kaleidoscope VR intervention group (Experimental): Children wore a virtual reality headset displaying a 3D kaleidoscope video with colorful geometric patterns. The headset was applied 2-3 minutes before peripheral intravenous catheterization and continued during the procedure to distract the child and reduce procedural pain and fear.
  Interventions: Device: Virtual Reality
- Routine care control group (No Intervention): Children received standard peripheral intravenous catheterization in the pediatric surgery unit without any additional distraction intervention.

INTERVENTIONS:
Device: Virtual Reality — 1. Aquarium VR Video (3D)
     Children in this group wore a virtual reality headset displaying a 3D Aquarium video. The video included underwater scenes with fish, sharks, and marine mammals. The VR headset was applied 2-3 minutes before the peripheral intravenous catheterization procedure and continued during the procedure to provide distraction.
  2. Kaleidoscope VR Video (3D)
     Children in this group wore a virtual reality headset displaying a 3D Kaleidoscope video consisting of colorful, shifting geometric patterns. The VR headset was applied 2-3 minutes before the peripheral intravenous catheterization procedure and continued during the procedure to distract the child and reduce procedural pain and fear.
  3. Routine Care (Control Group)
  Children in this group received standard peripheral intravenous catheterization procedure in the pediatric surgery unit without any additional distraction intervention.
  Arms: Aquarium VR intervention group; Kaleidoscope VR intervention group

SUMMARY:
This study aims to evaluate the effect of two different virtual reality (VR) applications on children's pain, fear, and physiological parameters during peripheral intravenous catheterization. Children between the ages of 7 and 12 who are scheduled for day surgery in the pediatric surgery unit will be randomly assigned to one of three groups: (1) Aquarium VR video, (2) Kaleidoscope VR video, or (3) routine care control group.

VR interventions will begin 2-3 minutes before the procedure and will continue throughout catheter insertion. The primary outcomes will include pain and fear levels measured by validated pediatric scales, while secondary outcomes will focus on physiological parameters such as heart rate, respiratory rate, body temperature, and oxygen saturation.

The purpose of this research is to determine whether distraction with VR technology can reduce procedural pain and fear in children, improve their cooperation during invasive procedures, and support atraumatic care practices in pediatric nursing.

DETAILED DESCRIPTION:
Children often experience pain, fear, and anxiety during invasive procedures such as peripheral intravenous catheterization. These negative experiences may reduce cooperation during treatment, cause long-term traumatic memories, and lower trust in health care. Non-pharmacological distraction methods have recently gained importance as safe, effective, and atraumatic strategies to reduce procedural pain in children. Virtual reality (VR) is a promising distraction tool that provides immersive visual and auditory stimuli, isolating the child from the hospital environment and redirecting attention away from the procedure.

This randomized controlled study will investigate the effect of two different VR applications-Aquarium VR video and Kaleidoscope VR video-on children's pain, fear, and physiological responses during peripheral intravenous catheterization. A total of 170 children, aged 7-12 years and scheduled for day surgery in the pediatric surgery unit, will be randomly assigned to one of three groups: Aquarium VR intervention, Kaleidoscope VR intervention, or routine care control. The VR interventions will start 2-3 minutes before the procedure and continue throughout catheter insertion.

Primary outcomes will be pain and fear levels, measured using validated pediatric scales including the Visual Analog Scale (VAS), Wong-Baker Faces Pain Rating Scale, and the Children's Fear Scale. Secondary outcomes will include physiological parameters (heart rate, respiratory rate, body temperature, and oxygen saturation) recorded before and after the procedure.

The study will provide evidence on whether distraction through VR can reduce pain and fear during intravenous catheterization in children and support atraumatic care principles in pediatric nursing. The findings may guide health professionals in adopting VR technology as a non-pharmacological intervention to improve the quality of care and enhance patient and family satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7-12 years
* Scheduled for day surgery in the pediatric surgery unit
* Undergoing first-time peripheral intravenous catheterization in the clinic
* Both child and parent provide informed consent/assent to participate
* Child and parent have no speech or visual impairment

Exclusion Criteria:

* Children younger than 7 or older than 12 years
* Not scheduled for day surgery in the pediatric surgery unit
* Child or parent declining participation
* Presence of speech or visual impairment in child or parent

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity during peripheral intravenous catheterization | Up to 10 minutes during and after the procedure.
  Pain intensity will be measured using the Visual Analog Scale (VAS), which is a 10 cm line anchored by "no pain" (0) and "worst possible pain" (10). Higher scores indicate greater pain intensity. Assessments will be made at baseline (before the procedure), during, and immediately after peripheral intravenous catheter insertion.
Pain intensity measured by Wong-Baker Faces Pain Rating Scale | Up to 10 minutes during and after peripheral intravenous catheterization.
  This scale ranges from 0 ("no hurt") to 5 ("hurts worst") with six faces representing increasing levels of pain. Higher scores indicate greater pain intensity.
Fear intensity measured by Children's Fear Scale (CFS) | Up to 10 minutes during and after peripheral intravenous catheterization.
  CFS consists of 5 faces scored from 0 (no fear) to 4 (highest fear). Higher scores indicate greater fear.

SECONDARY OUTCOMES:
Heart rate (beats per minute) | Immediately before and up to 10 minutes after the procedure.
  Heart rate will be recorded before and after peripheral intravenous catheterization. Changes in heart rate will be compared between groups.
Respiratory rate (breaths per minute) | Immediately before and up to 10 minutes after the procedure.
  Respiratory rate will be recorded before and after peripheral intravenous catheterization. Changes in respiratory rate will be compared between groups.
Blood pressure (systolic and diastolic mmHg) | Immediately before and up to 10 minutes after the procedure.
  Systolic and diastolic blood pressure will be recorded before and after peripheral intravenous catheterization. Changes in blood pressure will be compared between groups.
Oxygen saturation (percentage, %) | Immediately before and up to 10 minutes after the procedure.
  Peripheral oxygen saturation (SpO2) will be recorded before and after peripheral intravenous catheterization. Changes in oxygen saturation will be compared between groups.

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results of this study (text, tables, figures) will be made available upon reasonable request to the corresponding researcher after publication. Data will be shared with researchers who provide a methodologically sound proposal, and access will be granted through a data sharing agreement.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available beginning 6 months after publication and will be accessible for up to 5 years.
Access Criteria: Data will be shared with qualified researchers who submit a methodologically sound proposal and obtain approval from the principal investigator. Access will be granted through a data sharing agreement.